CLINICAL TRIAL: NCT03097432
Title: A Prospective, Open, Multi-centre, Non-interventional Study to Assess the Tolerability, the Safety Profile and the Adherence of Different Up-dosing Schemes for a Sublingual Immunotherapy Treatment
Brief Title: Non-interventional Study to Assess the Tolerability, the Safety Profile and the Adherence of Different Up-dosing Schemes for a Sublingual Immunotherapy Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: Bencard Allergie GmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ralph Mösges, Prof. Dr. med. Ralph Mösges, University Hospital of Cologne
Other Study IDs: Oralvac Compact Bäume
Record Dates: First submitted 2017-03-17; First posted 2017-03-31 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ORALVAC COMPACT BÄUME: This non-interventional study was initiated to document the up-dosing period of children and adults with allergic rhinoconjunctivitis and/or allergic asthma treated with a SLIT containing purified, aqueous extracts of birch, alder, and hazel pollen. The following up-dosing schemes were freely selectable: scheme A consists of an up-dosing period of 12 days at the patient´s home using the standardized pollen extract in three different solution strengths to reach the maximum dose; scheme B performed only with the highest solution strength at the physician's office within 2 hours; and the new scheme C which is a regimen for initiation at the physician's office and continuation at the patient's home also exclusively using the highest solution strength and takes 4 days.
  Interventions: Drug: ORALVAC COMPACT BÄUME

INTERVENTIONS:
Drug: ORALVAC COMPACT BÄUME

SUMMARY:
This prospective open multi-centre non-interventional study initiated to document the up-dosing period of children and adults with allergic rhinoconjunctivitis and/or allergic asthma treated with a SLIT containing purified, aqueous extracts of birch, alder, and hazel pollen. The following up-dosing schemes are freely selectable: scheme A consists of an up-dosing period of 12 days at the patient´s home using the standardized pollen extract in three different solution strengths to reach the maximum dose; scheme B is performed only with the highest solution strength at the physician's office within 2 hours; and the new scheme C which is a regimen for initiation at the physician's office and continuation at the patient's home also exclusively using the highest solution strength and takes 4 days. Data are documented by physicians and in patients´ diaries.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the age of 2 years and older suffering from a tree pollen induced seasonal allergic rhinitis

Exclusion Criteria:

* Patients suffering from acute or chronic infections or inflammations
* Patients suffering from secondary modifications of the target organ with function impairment (emphysema, bronchiectasis)
* Patients suffering from severe and uncontrolled asthma
* Patients with a known severe autoimmune disease
* Patients with active malignant disease
* Patients requiring beta-blockers
* Patients having any contraindication for the use of adrenaline
* Patients with a hypersensitivity to the excipients of the drug

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults, adolescents and children from the age of 2 on, who suffer from seasonal allergic rhinoconjunctivitis causued by tree pollen.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and Tolerability) | up to 12 days of the up-dosing phase
  Tolerability and safety will be assessed by the frequency and intensity of local reactions (mouth, lips, pharynx/throat, gastrointestinal tract) and systemic reactions (skin, airways, others) during the up-dosing phase.
Improvement of rhinoconjunctivitis symptoms and intake of rescue medication (efficacy) | through study completion, tree pollen season 2017
  Efficacy will be assessed by the improvement of rhinoconjunctivitis symptoms and intake of rescue medication during the tree pollen season 2017

SECONDARY OUTCOMES:
Evaluation of tolerability and safety | up to 12 days of the up-dosing phase
  Tolerability and safety of the treatment with ORALVAC COMPACT BÄUME will be evaluated by the frequency and intensity of miscellaneous adverse events during the up-dosing phase.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kramer, Prof. Dr., Study Director — Bencard Allergie GmbH
Locations (1):
- UHCologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mosges R, Breitruck NY, Allekotte S, Shah-Hosseini K, Dao VA, Zieglmayer P, Birkholz K, Hess M, Bastl M, Bastl K, Berger U, Kramer MF, Guethoff S. Shortened up-dosing with sublingual immunotherapy drops containing tree allergens is well tolerated and elicits dose-dependent clinical effects during the first pollen season. World Allergy Organ J. 2019 Mar 8;12(2):100012. doi: 10.1016/j.waojou.2019.100012. eCollection 2019. PMID 30937138